CLINICAL TRIAL: NCT02607761
Title: Fertility Awareness in University Students
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Mariana Veloso Martins, Mariana Veloso Martins, PhD, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FPCEUP/RH1; PTDC/MHC-PSC/4195/2012 (Other Grant/Funding Number: Portuguese Foundation for Science and Technology)
Record Dates: First submitted 2015-10-15; First posted 2015-11-18 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Educational Video
Keywords: infertility; fertility awareness; health interventions; young adults
MeSH Terms: conditions — Infertility | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention Group (Experimental): 2 minutes video with information and images on age-related fertility, infertility definitions, infertility risk factors, probabilities of fecundity according to age and cycle.
  Interventions: Other: Video
- Control (No Intervention): No intervention
- Control 1 (Active Comparator): 2 minutes video with same images but information on work-family balance.
  Interventions: Other: Video

INTERVENTIONS:
Other: Video — Video-Audio Media
  Arms: Control 1; Intervention Group

SUMMARY:
Recent evidence showed that undergraduate students have inappropriate knowledge about reproductive health and infertility.

The investigators' aim was to assess the effectiveness of a brief intervention (video) in increasing the knowledge regarding fertility issues, fertility risk factors and infertility definition.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate student

Exclusion Criteria:

* Having knowledge of a fertility problem

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 323 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
change in fertility knowledge | T1 - immediatly after intervention; T2 - one week later; T3 - one month later; T4 - 12 months later
  This measure assesses fertility knowledge by asking 10 questions on the probability of conception and fertility treatment success rates.

SECONDARY OUTCOMES:
change in age of desired parenthood | T1 - immediatly after intervention; T2 - one week later; T3 - one month later; T4 - 12 months later
  Subjects are asked to write how many children would they like to have in the future and what is the desired age for having the first and the last child.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Porto, Faculty of Psychology and Educational and Education Sciences, Porto, Porto District, Portugal

REFERENCES:
- [Derived] Conceicao C, Pedro J, Martins MV. Effectiveness of a video intervention on fertility knowledge among university students: a randomised pre-test/post-test study. Eur J Contracept Reprod Health Care. 2017 Apr;22(2):107-113. doi: 10.1080/13625187.2017.1288903. Epub 2017 Feb 14. PMID 28256912